CLINICAL TRIAL: NCT00731679
Title: A Phase 3, Randomized, Double-blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of Rifaximin 550 mg TID in the Treatment of Subjects With Non-Constipation Irritable Bowel Syndrome
Brief Title: Rifaximin 3 Times/Day (TID) for Non-Constipation Irritable Bowel Syndrome (IBS)
Acronym: TARGET 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RFIB3007
Record Dates: First submitted 2008-07-16; First posted 2008-08-11 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Non-Constipation Irritable Bowel Syndrome
Keywords: IBS; Abdominal pain; Bloating; Diarrhea; Rifaximin
MeSH Terms: conditions — Abdominal Pain; Diarrhea | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects received placebo tablets 3 times daily for 2 weeks and were followed for 10 weeks after completion of the treatment period.
  Interventions: Drug: Placebo
- Rifaximin (Experimental): Subjects received rifaximin 550 mg tablets 3 times daily for 2 weeks and were followed for 10 weeks after completion of the treatment period.
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin
  Arms: Rifaximin
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of a 14-day course of rifaximin given 3 times a day vs. placebo in providing adequate relief of IBS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed IBS diagnosis per Rome II for diagnosis of IBS.
* Colonoscopy within 2 years as part of IBS diagnostic evaluation.
* Has active symptoms of non-constipation IBS at baseline as measured by average daily scores for abdominal pain/discomfort, bloating, and stool consistency.

Exclusion Criteria:

* Symptoms of constipation.
* History of other gastrointestinal diseases.
* Type 1 or 2 diabetes.
* Lactose intolerance not controlled by lactose-free diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enoch Bortey, Study Director — Bausch Health Americas, Inc.
Locations (88):
- United States (81):
  - Hueytown, Alabama
  - Phoenix, Arizona
  - Sierra Vista, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Sherwood, Arkansas
  - Anaheim, California
  - Lancaster, California
  - Los Angeles, California
  - Murrieta, California
  - San Diego, California
  - Lakewood, Colorado
  - Bridgeport, Connecticut
  - Torrington, Connecticut
  - Altamonte Springs, Florida
  - Boynton Beach, Florida
  - Gainesville, Florida
  - Hollywood, Florida
  - Jupiter, Florida
  - Lauderdale Lakes, Florida
  - Maitland, Florida
  - Naples, Florida
  - New Port Richey, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Winter Garden, Florida
  - Winter Park, Florida
  - Topeka, Kansas
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Hagerstown, Maryland
  - Silver Spring, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Paw Paw, Michigan
  - Jackson, Mississippi
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Elizabeth, New Jersey
  - Lumberton, New Jersey
  - Bayside, New York
  - Brooklyn, New York
  - New York, New York
  - Troy, New York
  - Asheboro, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Fayetteville, North Carolina
  - Greensboro, North Carolina
  - High Point, North Carolina
  - Mooresville, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Zanesville, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Lancaster, Pennsylvania
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Johnson City, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Pasadena, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Ogden, Utah
  - West Jordan, Utah
  - Chesapeake, Virginia
  - Lynchburg, Virginia
  - Bellevue, Washington
  - Spokane, Washington
  - West Bend, Wisconsin
- Canada (7):
  - St. John's, Newfoundland and Labrador
  - Corunna, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Niagara Falls, Ontario
  - Sarnia, Ontario

REFERENCES:
- [Result] Pimentel M, Lembo A, Chey WD, Zakko S, Ringel Y, Yu J, Mareya SM, Shaw AL, Bortey E, Forbes WP; TARGET Study Group. Rifaximin therapy for patients with irritable bowel syndrome without constipation. N Engl J Med. 2011 Jan 6;364(1):22-32. doi: 10.1056/NEJMoa1004409. PMID 21208106
- [Derived] Lacy BE, Chang L, Rao SSC, Heimanson Z, Sayuk GS. Rifaximin Treatment for Individual and Multiple Symptoms of Irritable Bowel Syndrome With Diarrhea: An Analysis Using New End Points. Clin Ther. 2023 Mar;45(3):198-209. doi: 10.1016/j.clinthera.2023.01.010. Epub 2023 Mar 14. PMID 36922331
- [Derived] Schoenfeld P, Pimentel M, Chang L, Lembo A, Chey WD, Yu J, Paterson C, Bortey E, Forbes WP. Safety and tolerability of rifaximin for the treatment of irritable bowel syndrome without constipation: a pooled analysis of randomised, double-blind, placebo-controlled trials. Aliment Pharmacol Ther. 2014 May;39(10):1161-8. doi: 10.1111/apt.12735. Epub 2014 Apr 3. PMID 24697851

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Rifaximin
Started | 314 | 309
Completed | 292 | 283
Not Completed | 22 | 26
Not completed — Adverse Event | 7 | 8
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Lost to Follow-up | 7 | 8
Not completed — Noncompliance | 0 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population was the intent-to-treat population, defined as subjects who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rifaximin | Total
Number analyzed (Participants) | 314 | 309 | 623
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 275 | 274 | 549
  >=65 years | 38 | 34 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (14.6) | 46.2 (15.0) | 45.8 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 235 | 457
  Male | 92 | 74 | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 30 | 24 | 54
  White | 280 | 281 | 561
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Had Adequate Relief of Global IBS Symptoms for at Least 2 of the 4 Weeks During the Primary Evaluation Period (ie, Weeks 3 Through 6).
Description: The primary outcome measure is assessed during the 4-week period (ie, Weeks 3 through 6) immediately following 2 weeks of treatment with study drug. Adequate relief of global IBS symptoms was defined as a response of "yes" to the following question, which was asked weekly (every 7 days): "In regard to all your symptoms of IBS, as compared to the way you felt before you started study medication, have you, in the past 7 days, had adequate relief of your IBS symptoms? [Yes/No]"
Time Frame: 4 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | Rifaximin
Number analyzed (Participants) | 314 | 309
percentage of responders | 31.2 | 40.8
Statistical Analysis 1: Comparison: Placebo vs Rifaximin; Test type: Superiority or Other; p = 0.01, Regression, Logistic; The p-value was obtained from a logistic regression model with fixed effects for treatment arm and analysis center

2. Secondary Outcome: Proportion of Subjects Who Had Adequate Relief of IBS-related Bloating for at Least 2 of the 4 Weeks During the Primary Evaluation Period (ie, Weeks 3 Through 6).
Description: The secondary outcome measure is assessed during the 4-week period (ie, Weeks 3 through 6) immediately following 2 weeks of treatment with study drug. Adequate relief of bloating was defined as a response of "yes" to the following question, which was asked weekly (every 7 days): "In regard to your symptom of bloating, as compared to the way you felt before you started study medication, have you, in the past 7 days, had adequate relief of your IBS symptom of bloating? [Yes/No]."
Time Frame: 4 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | Rifaximin
Number analyzed (Participants) | 314 | 309
percentage of responders | 28.7 | 39.5
Statistical Analysis 1: Comparison: Placebo vs Rifaximin; Test type: Superiority or Other; p = 0.005, Regression, Logistic; The p-value was obtained from a logistic regression model with fixed effects for treatment arm and analysis center

ADVERSE EVENTS:
Time Frame: 12 weeks. Adverse events were collected during the 2-week treatment period and during the 10-week follow-up period.
Description: Non-systematic (patient reports) and systematic methods (investigator examinations/laboratory tests) were used to collect adverse events. A subject reporting more than one adverse event for a particular MedDRA preferred term or system organ class was counted only once for that MedDRA preferred term or system organ class.
Arm/Group | Placebo | Rifaximin
Serious Adverse Events (participants affected / at risk) | 8/314 | 3/309
Other Adverse Events (participants affected / at risk) | 101/314 | 103/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=314) | Rifaximin (N=309)
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0
Labile hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=314) | Rifaximin (N=309)
Abdominal distension (Gastrointestinal disorders) | 7 | 7
Abdominal pain (Gastrointestinal disorders) | 23 | 19
Diarrhoea (Gastrointestinal disorders) | 15 | 14
Flatulence (Gastrointestinal disorders) | 11 | 6
Nausea (Gastrointestinal disorders) | 13 | 22
Vomiting (Gastrointestinal disorders) | 8 | 11
Bronchitis (Infections and infestations) | 8 | 6
Nasopharyngitis (Infections and infestations) | 18 | 7
Sinusitis (Infections and infestations) | 12 | 7
Upper respiratory tract infection (Infections and infestations) | 9 | 8
Urinary tract infection (Infections and infestations) | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Headache (Nervous system disorders) | 16 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days